CLINICAL TRIAL: NCT03360136
Title: Multiprofessional Rehabilitation for Exhaustion Disorder
Brief Title: Open Clinical Trial of CBT-based Multiprofessional Rehabilitation for Exhaustion Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: PBM Sweden AB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1834- 31/2
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Exhaustion; Syndrome; Burnout, Professional; Burnout Syndrome; Adjustment Disorders
Keywords: Exhaustion Disorder; Burnout; Clinical Burnout
MeSH Terms: conditions — Syndrome; Burnout, Professional; Burnout, Psychological; Adjustment Disorders

STUDY DESIGN:
Intervention Model Description: Open Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-professional CBT-rehabilitation (Other): 24 weeks CBT-based multi-professional rehabilitation.
  Interventions: Behavioral: Multi-professional CBT-rehabilitation

INTERVENTIONS:
Behavioral: Multi-professional CBT-rehabilitation — See "Detailed description"

SUMMARY:
Stress-related mental disorders are today the leading cause of long-term sick leave in Sweden, and a large part of this increase is due to Clinical burnout, in Sweden called "Exhaustion disorder" (ED). Even though clinical guidelines recommend multi-professional rehabilitation (MPR) for ED, few studies have evaluated the effects of these treatment programs in clinical practice. This large-scale open clinical trial investigates whether MPR for ED seems to alleviate symptoms of ED and if it results in return-to-work.

DETAILED DESCRIPTION:
This study is carried out at two specialized stress rehabilitation centers in Stockholm. All patients included in the clinics stress rehabilitation program are asked to participate in the study and are recruited consecutively from October 2017 throughout December 2018. An estimate of 400 patients will be included. The treatment program is a 24-week Multiprofessional standardized CBT-rehabilitation consisting of a nine-session CBT group treatment (stress management) followed by a seven-session group treatment in applied relaxation. Parallel to the group treatments patients receives nine sessions of individual CBT, three visits to an MD (for medication, follow-up, and sick-listing), two individual sessions to a physiotherapist and a three session-exercise group. Also, vocational measures are taken through rehabilitation meetings together with the patient's employer (if an employer exists). Primary treatment outcomes will be return-to-work (RTW) and symptoms of ED, anxiety, and depression. Secondary treatment outcomes will be quality of life, pathological worry, psychological flexibility, clinical perfectionism, insomnia, burnout, and symptoms. Predictors of symptom development and RTW will be explored. Also, comorbidity of chronic pain, negative effects of psychotherapy and treatment credibility will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed exhaustion disorder according to criteria established by the Swedish National Board of Health and Welfare
* 18 - 64 years of age
* Considered suitable for multimodal rehabilitation in group
* Self-rating of > 4,5 på SMBQ

Exclusion Criteria:

* Abuse of alcohol or drugs
* Moderate-high suicidal risk
* Severe psychiatric illness (severe depression, bipolar, schizophrenia etc.)
* Untreated PTSD

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exhaustion symptoms | Week 12 and 24
  Self-reported change in Karolinska Exhaustion Disorder Scale, 9 items
Change from baseline to follow-up in exhaustion symptoms | Week 12, 24 and 76
  Self-reported change in Karolinska Exhaustion Disorder Scale, 9 items
Change from baseline in depression | Week 12 and 24
  Self-reported change in Hospital Anxiety Depressin Scale (HADS), 14 items
Change from baseline to follow-up in depression | Week 12, 24 and 76
  Self-reported change in Hospital Anxiety Depressin Scale (HADS), 14 items
Change from baseline in anxiety | Week 12 and 24
  Self-reported change in Hospital Anxiety Depressin Scale (HADS), 14 items
Change from baseline to follow-up in anxiety | Week 12, 24 and 76
  Self-reported change in Hospital Anxiety Depressin Scale (HADS), 14 items
Change from baseline in employment rate | Week 24
  Sick-leave data collected from the Swedish Social Insurance Agency
Change from baseline to follow-up in employment rate | Week 24 and 76
  Sick-leave data collected from the Swedish Social Insurance Agency

SECONDARY OUTCOMES:
Change from baseline in Quality of life | Week 24
  Self-reported change in EQ5D, 5 items
Change from baseline to follow-up in Quality of life | Week 24 and 76
  Self-reported change in EQ5D, 5 items
Change from baseline in insomnia symptoms | Week 12 and 24
  Self-reported change in Insomnia Severity Index (ISI), 7 items
Change from baseline to follow-up in insomnia symptoms | Week 12, 24 and 76
  Self-reported change in Insomnia Severity Index (ISI), 7 items
Change from baseline in Clinical Perfectionism | Week 12 and 24
  Self-reported change in Clinical Perfectionism Questionnaire (CPQ), 12 items
Change from baseline to follow-up in Clinical Perfectionism | Week 12, 24 and 76
  Self-reported change in Clinical Perfectionism Questionnaire (CPQ), 12 items
Change from baseline in Psychological Flexibility | Week 12 and 24
  Self-reported change in the Swedish Acceptance and Action Questionnaire (SAAQ), 6 items
Change from baseline to follow-up in Psychological Flexibility | Week 12, 24 and 76
  Self-reported change in the Swedish Acceptance and Action Questionnaire (SAAQ), 6 items
Change from baseline in pathological worry | Week 12 and 24
  Self reported change in Penn State Worry Questionnaire ultra-brief (PSWQ-brief), 3 items
Change from baseline to follow-up in pathological worry | Week 12, 24 and 76
  Self reported change in Penn State Worry Questionnaire ultra-brief (PSWQ-brief), 3 items
Change from baseline in perceived work ability | Week 12 and 24
  Self-rated work ability, 1 single item from Work Ability index (WAI)
Change from baseline to follow up in perceived work ability | Week 12, 24 and 76
  Self-rated work ability, 1 single item from Work Ability index (WAI)
Change from baseline in burnout | Week 12 and 24
  Self-rated burnout in Shirom Melamed Burnout Questionnaire (SMBQ), 22 items
Change from baseline to follow-up in burnout | Week 12, 24 and 76
  Self-rated burnout in Shirom Melamed Burnout Questionnaire (SMBQ), 22 items

OTHER OUTCOMES:
Negative Effects of psychotherapy | at 24 week only
  Self-Reported negative effects in Negative Effects Questionnaire, 32 items
Treatment credibility rating | Baseline and at 12 weeks
  Self-reported treatment credibility, treatment Credibility Scale (TCS), 5 items

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Brodda Jansen, Assoc. Proff., Study Chair — Karolinska University
Locations (2):
- Sweden (2):
  - PBM Sweden AB Globen, Stockholm, Södermanland County
  - PBM Sweden City, Stockholm, Uppland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martensson G, Johansson F, Buhrman M, Ahs F, Clason van de Leur J. A network analysis of exhaustion disorder symptoms throughout treatment. BMC Psychiatry. 2024 May 23;24(1):389. doi: 10.1186/s12888-024-05842-9. PMID 38783205
- [Derived] van de Leur JC, Buhrman M, Wallby K, Karlstrom A, Johansson F. Associations between improvements in psychological variables and subsequent sick leave among persons receiving a multimodal intervention for exhaustion disorder. BMC Public Health. 2023 Oct 11;23(1):1976. doi: 10.1186/s12889-023-16799-x. PMID 37821913
- [Derived] van de Leur JC, Buhrman M, Ahs F, Rozental A, Jansen GB. Standardized multimodal intervention for stress-induced exhaustion disorder: an open trial in a clinical setting. BMC Psychiatry. 2020 Nov 5;20(1):526. doi: 10.1186/s12888-020-02907-3. PMID 33153461